CLINICAL TRIAL: NCT01250678
Title: Neurocognitive Changes in Patients With Remitting Relapsing Multiple Sclerosis Treated With Natalizumab
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: Biogen (Industry)
Responsible Party: Murat YIldiz, Cantonal Hospital Saint Gallen
Other Study IDs: CogNtz
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
Keywords: multiple sclerosis; cognitive impairment; natalizumab; SDMT
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- neurocognitive impaired: MS patients treated with natalizumab who at the beginning of the study suffer from cognitive impairment
- neurocognitive non-impaired: MS patients treated with natalizumab who at the beginning of the study do not suffer from cognitive impairment

SUMMARY:
Cognitive impairment is seen in about half of patients with relapsing remitting MS. Our knowledge about long term development of cognitive performance under natalizumab therapy is limited. We want to demonstrate with this study that patients treated with ntz improve in neurocognitive tests over the long term.

DETAILED DESCRIPTION:
Impaired cognitive function may represent damage to brain regions that are not involved in physical functions, hence may not be detected during routine neurological assessment. Despite the high prevalence of cognitive impairment in MS, cognitive function is not assessed routinely in clinical practice. The perception that cognitive assessments are costly, time-consuming, complicated, and difficult to administer and interpret has contributed, at least in part, to the failure to incorporate cognitive testing into standard clinical evaluation of patients with MS.

Cognitive impairment may also reduce the ability of patients to comprehend and adhere to treatment concepts (Bobholz 2003). Early detection of cognitive impairment is important to initiate therapeutic intervention, even though the optimal treatment of cognitive decline in MS is at the moment controversial.

Preliminary studies suggest an essential role of disease modifying therapies (DMT) in inhibition of cognitive deterioration in patients with MS (Barak 2002, Flechter 2007). Data about long term cognitive performance of multiple sclerosis patients treated with natalizumab is limited. One study demonstrated in MS patients treated with natalizumab an improvement in SDMT (Symbol Digit Modalities Test) of 16.4% over a period of 2 years (Piehl 2010). SDMT is a screening tool for cognitive impairment in MS patients, mainly measuring working memory and speed processing. As SDMT only covers a part of the neurocognitive impairments seen in MS patients, there is a need for further studies to gain a more complete picture.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 55 years at presentation
* Diagnosis of relapsing-remitting MS according to revised McDonald criteria 2005
* Patients treated with ntz
* EDSS under 5.5

Exclusion Criteria:

* Brain pathology other than MS
* Known history of head trauma
* Pure spinal manifestation of demyelization
* Neuromyelitis optica
* Primary and secondary progressive MS
* Benzodiazepine intake within the last three months
* Relapse within the last three months
* Steroid intake within the last three months
* History of severe depressive disorder and/or suicidality, seizure, drug or alcohol abuse
* No informed consent
* Insufficient knowledge of German

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MS-patients will be recruited in the outpatient clinic of the neurology department of the cantonal hospital of Saint Gallen, responsible for treatment of MS patients of Northeast Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The Symbol Digit Modalities Test (SDMT) | 3 years
  SDMT is an easily administered brief screening tool for cognitive dysfunction in MS. Patients view a key presenting nine numbers paired with symbols. Below the key is an array of symbols paired with empty spaces, the patient's task being to voice the matching number for each symbol as rapidly as possible.

SECONDARY OUTCOMES:
Multiple Sclerosis Inventory Cognition (MUSIC) | 3 years
  MUSIC is a cognitive screening instrument. It assesses the cognitive core deficit in MS: mental flexibility, attention, information processing speed, memory and inhibitory control and includes also 3 items derived from a factorial analysis to examine cognitive, motor and psychosocial fatigue, respectively.
TAP subtest Alertness | 3 years
  TAP subtest Alertness measures the subject's ability to respond to a visual stimulus and to increase the attentional level in expectance of a stimulus of high priority. The computer-assisted test is given under 2 conditions: Simple reaction time to a visual stimulus (Greek cross) appearing at randomly varying intervals on the monitor screen is measured. In the second condition, the visual stimulus (= critical stimulus) is preceded by a cue sound presented as warning tone.
Composite neurocognitive index | 3 years
  Overall neurocognitive status will be assessed with a composite cognitive index score representing the sum of the scores for the individual tests: TAP subtest Alertness, MUSIC and SDMT.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yildiz, MD, Principal Investigator — Cantonal Hospital Saint Gallen
Locations (1):
- Cantonal Hospital of Saint Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] Yildiz M, Tettenborn B, Radue EW, Bendfeldt K, Borgwardt S. Association of cognitive impairment and lesion volumes in multiple sclerosis--a MRI study. Clin Neurol Neurosurg. 2014 Dec;127:54-8. doi: 10.1016/j.clineuro.2014.09.019. Epub 2014 Oct 14. PMID 25459243